CLINICAL TRIAL: NCT03498456
Title: A Phase 3, Randomized, Double-blind, Active-controlled, Multicenter Study to Evaluate the Efficacy and Safety of a Triple Therapy With Tegoprazan, Amoxicillin, and Clarithromycin in H. Pylori Positive Patients
Brief Title: Triple Therapy With Tegoprazan in H. Pylori Positive Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CJ_APA_307
Record Dates: First submitted 2018-04-08; First posted 2018-04-13 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Helicobacter Pylori Infection
MeSH Terms: interventions — tegoprazan; Lansoprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tegoprazan/Amoxicillin/Clarithromycin (Experimental): Tegoprazan 50 mg / Amoxicillin 1000 mg / Clarithromycin 500 mg
  Interventions: Drug: Tegoprazan/Amoxicillin/Clarithromycin
- Lansoprazole/Amoxicillin/Clarithromycin (Active Comparator): Lansoprazole 30 mg / Amoxicillin 1000 mg / Clarithromycin 500 mg
  Interventions: Drug: Lansoprazole/Amoxicillin/Clarithromycin

INTERVENTIONS:
Drug: Tegoprazan/Amoxicillin/Clarithromycin — Tegoprazan 50 mg + Amoxicillin 1000 mg + Clarithromycin 500 mg bid. This therapy will be administered for a total of 7 days, in fasting conditions in the morning and the evening.
  Other Names: Tegoprazan triple therapy (TAC)
  Arms: Tegoprazan/Amoxicillin/Clarithromycin
Drug: Lansoprazole/Amoxicillin/Clarithromycin — Lansoprazole 30 mg + Amoxicillin 1000 mg + Clarithromycin 500 mg bid. This therapy will be administered for a total of 7 days, in fasting conditions in the morning and the evening.
  Other Names: Lansoprazole triple therapy (LAC)
  Arms: Lansoprazole/Amoxicillin/Clarithromycin

SUMMARY:
The current study is designed to demonstrate the non-inferiority of tegoprazan triple therapy (tegoprazan, amoxicillin, and clarithromycin; hereinafter TAC) to lansoprazole triple therapy (lansoprazole, amoxicillin, and clarithromycin; hereinafter LAC) in terms of H. pylori eradication rate and to evaluate the safety of tegoprazan after oral administration of the therapy for 7 days, twice daily in H. pylori positive patients.

DETAILED DESCRIPTION:
This is a randomized, double blind, active controlled, multicenter, Phase 3 study to demonstrate the non-inferiority of tegoprazan triple therapy (TAC) to lansoprazole triple therapy (LAC) in terms of H. pylori eradication rate and to evaluate the safety of tegoprazan in H. pylori positive patients after oral administration of therapy for 7 days, twice daily. After the treatment, UBT test will be conducted to confirm the Helicobacter pylori eradication.

ELIGIBILITY:
Inclusion Criteria:

* H. pylori positive based on the screening test
* Peptic ulcer disease

Exclusion Criteria:

* Prior treatment for H. pylori eradication
* Prior use of proton pump inhibitors (PPIs), H2 receptor blockers, at a full dosage within 14 days
* Prior use of H. pylori eradication effective antibiotics, bismuth within 14 days

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 2018-06-28 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
H. pylori eradication rate | 6 weeks
  Subjects will be considered to succeed in achieving H. pylori eradication if subjects's negative UBT test.

CONTACTS AND LOCATIONS:
Overall Officials: Hwoon Yong Jung, Professor, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided